CLINICAL TRIAL: NCT03214367
Title: A Prospective, Randomized, Double-Blind Comparison of LY900014 to Insulin Lispro With an Open-Label Postprandial LY900014 Treatment Group, in Combination With Insulin Glargine or Insulin Degludec, in Adults With Type 1 Diabetes PRONTO-T1D
Brief Title: A Study of LY900014 in Participants With Type 1 Diabetes
Acronym: PRONTO-T1D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16313; I8B-MC-ITRM (Other: Eli Lilly and Company); 2015-005356-99 (EudraCT Number)
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin Glargine; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY900014 (Experimental): LY900014 given subcutaneously (SC) 0-2 minutes before each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
  Interventions: Drug: LY900014; Drug: Insulin Glargine; Drug: Insulin Degludec
- Insulin Lispro (Humalog) (Active Comparator): Insulin lispro given SC 0-2 minutes before each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
  Interventions: Drug: Insulin Lispro; Drug: Insulin Glargine; Drug: Insulin Degludec
- LY900014 Postmeal (Open Label) (Experimental): LY900014 given SC 20 minutes after the start of each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Prandial insulin doses were individualized and titrated according to protocol-defined targets.
  Interventions: Drug: LY900014; Drug: Insulin Glargine; Drug: Insulin Degludec
- LY900014 - Maximum Extended Enrollment (MEE) (Experimental): LY900014 given subcutaneously (SC) 0-2 minutes before each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
  Interventions: Drug: LY900014; Drug: Insulin Glargine; Drug: Insulin Degludec
- Insulin Lispro (Humalog)-MEE (Active Comparator): Insulin lispro given SC 0-2 minutes before each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
  Interventions: Drug: Insulin Lispro; Drug: Insulin Glargine; Drug: Insulin Degludec
- LY900014 Postmeal (Open Label)-MEE (Experimental): LY900014 given SC 20 minutes after the start of each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Prandial insulin doses were individualized and titrated according to protocol-defined targets.
  Interventions: Drug: LY900014; Drug: Insulin Glargine; Drug: Insulin Degludec

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014; LY900014 - Maximum Extended Enrollment (MEE); LY900014 Postmeal (Open Label); LY900014 Postmeal (Open Label)-MEE
Drug: Insulin Lispro — Administered SC
  Other Names: Humalog
  Arms: Insulin Lispro (Humalog); Insulin Lispro (Humalog)-MEE
Drug: Insulin Glargine — Administered SC
Drug: Insulin Degludec — Administered SC

SUMMARY:
The main purpose of this study is to evaluate the efficacy of the study drug LY900014 compared to insulin lispro, both in combination with insulin glargine or insulin degludec, in adults with type 1 diabetes (T1D).

ELIGIBILITY:
Inclusion Criteria:

* Have T1D for at least 1 year prior to screening and continuously using insulin for at least 1 year.
* HbA1c of ≥7.0 and ≤9.5%.
* Use insulin lispro, insulin aspart, or insulin glulisine as prandial insulin.
* Use insulin glargine, insulin detemir, insulin degludec, or neutral protamine Hagedorn (NPH) insulin as basal insulin.

Exclusion Criteria:

* Have used other antihyperglycemic medications or therapies (inhaled, oral or injectable) within 90-days of screening.
* Have had more than 1 severe hypoglycemic episode within 6 months of screening.
* Have had more than 1 hospitalization related to hyperglycemia or diabetic ketoacidosis within 6 months of screening.
* Have clinically significant gastrointestinal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1392 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (157):
- United States (43):
  - Internal Medicine Center LLC, Mobile, Alabama
  - John Muir Physician Network Clinical Research Center, Concord, California
  - AMCR Institute INC, Escondido, California
  - Valley Endocrine, Fresno, Fresno, California
  - Marin Endocrine Associates, Greenbrae, California
  - Diabetes and Endocrine Associates, La Mesa, California
  - University Clinical Investigators, Inc., Tustin, California
  - Coastal Metabolic Research Centre, Ventura, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - The Center For Diabetes & Endocrine Care, Fort Lauderdale, Florida
  - East Coast Institute For Research, Jacksonville, Florida
  - Sun Coast Clinical Research, Inc, New Port Richey, Florida
  - Metabolic Research Institute Inc., West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - East Coast Institute For Research, Macon, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - East West Medical Institute, Honolulu, Hawaii
  - Northwest Clinical Trials, Boise, Idaho
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Iderc, P.L.C., West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cotton O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - MassResearch, Waltham, Massachusetts
  - Palm Research Center, Las Vegas, Nevada
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - Manhattan Medical Research, New York, New York
  - Physicians East, Greenville, North Carolina
  - Diabetes & Endocrinology Consultants PC, Morehead City, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Your Diabetes Endocrine Nutrition Group PC, Mentor, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Partners in Nephrology & Endocrinology, Pittsburgh, Pennsylvania
  - Sudir Bansal M.D. Inc., Warwick, Rhode Island
  - University Diabetes and Endocrine Consultants, Chattanooga, Tennessee
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Texas Diabetes and Endocrinology, P.A., Round Rock, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Progressive Clinical Research, Bountiful, Utah
  - Private: Dr. Larry Stonesifer, Federal Way, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Argentina (7):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Caba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Autonoma de Buenos Aire
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ciudad Autonoma de Buenos Aire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Box Hill
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Geelong
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Merewether
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Oaklands Park
- Austria (3):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Vienna
- For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., São Paulo, Brazil
- Germany (10):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Bad Mergentheim
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Falkensee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Hessen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Magdeburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mayen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oldenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rheine
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Saterland
- Greece (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ampelokipoi
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Larissa
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Thermi
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Thessaloniki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- India (7):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Hyderabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indore
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Pune
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Secunderabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Visakhapatnam
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ravenna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siena
- Japan (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amagasaki
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Kamakura
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Miyazaki
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Naka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōsaka
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ōsaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Sasebo
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Shinjuku
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Mexico (4):
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zapopan
- New Zealand (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Takapuna, Auckland
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Auckland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Christchurch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellington
- Poland (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ruda Śląska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Puerto Rico (5):
  - Dr Altagracia Aurora Alcantara Gonzalez, Bayamón
  - Advanced Clinical Research, LLC, Bayamón
  - Manati Center for Clinical Research Inc, Manatí
  - Martha Gomez Cuellar M.D., San Juan
  - Centro de Endocrinologia del Este, Yabucoa
- Romania (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bacau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lasi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ploieşti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Satu Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara
- Russia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kursk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
- Slovakia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Košice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malacky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nové Mesto nad Váhom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rožňava
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell, Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira, Valencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teruel
- Sweden (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Linköping
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
- Taiwan (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chang-hua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yongkang District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Piras de Oliveira C, Dellva MA, Bue-Valleskey J, Chang AM, Liao B. Fasting and postprandial plasma glucose contributions to hemoglobin A1c and time in range in people with diabetes on multiple daily injection insulin therapy: Results from the PRONTO-T1D and PRONTO-T2D clinical trials. J Diabetes Complications. 2024 Jan;38(1):108648. doi: 10.1016/j.jdiacomp.2023.108648. Epub 2023 Nov 16. PMID 38035641
- [Derived] Miura J, Nishiyama H, Imori M. Long-term Efficacy and Safety of Ultra Rapid Lispro in Japanese Patients With Type 1 Diabetes: Subpopulation Analysis of the 52-Week PRONTO-T1D Study. Diabetes Ther. 2021 Sep;12(9):2471-2484. doi: 10.1007/s13300-021-01124-9. Epub 2021 Aug 4. PMID 34347267
- [Derived] Bue-Valleskey J, Klaff L, Cho JI, Dellva MA, Schloot NC, Tobian J, Miura J, Dahl D. Long-Term Efficacy and Safety of Ultra Rapid Lispro (URLi) in Adults with Type 1 Diabetes: The PRONTO-T1D Extension. Diabetes Ther. 2021 Feb;12(2):569-580. doi: 10.1007/s13300-020-00987-8. Epub 2021 Jan 17. PMID 33458803
- [Derived] Miura J, Imori M, Nishiyama H, Imaoka T. Ultra-Rapid Lispro Efficacy and Safety Compared to Humalog(R) in Japanese Patients with Type 1 Diabetes: PRONTO-T1D Subpopulation Analysis. Diabetes Ther. 2020 Sep;11(9):2089-2104. doi: 10.1007/s13300-020-00892-0. Epub 2020 Jul 29. PMID 32728832
- See also: A Study of LY900014 in Participants With Type 1 Diabetes (PRONTO-T1D) — https://www.lillytrialguide.com/en-US/studies/type-1-diabetes/ITRM#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consists of 2 double-blind arms (LY900014 and Insulin Lispro (Humalog)) and one Open-label treatment group (LY900014 Postmeal).
  Double-blind group: The study included 8-week lead-in period followed by a 52-week treatment period.
  Open-label treatment group: The treatment period ended after 26 weeks.
Pre-assignment Details: The purpose of the Lead-in Period was to titrate basal insulin prior to randomization. Participants were then randomized to either LY900014 at mealtime, Insulin Lispro (Humalog) at mealtime, or LY900014 administered 20 minutes after the start of a meal (LY900014 Postmeal) in the treatment period (Period 2).
Groups:
- Insulin Lispro (Humalog) Lead-in: 100 units per milliliter (U/mL) Insulin lispro given subcutaneously (SC) 0-2 minutes before each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
- Insulin Lispro (Humalog); Insulin Lispro (Humalog) Lead-In Maximum Extended Enrollment; Insulin Lispro (Humalog)- Maximum Extended Enrollment (MEE): 100 U/mL Insulin lispro given subcutaneously (SC) 0-2 minutes before each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
- LY900014; LY900014-MEE: 100 U/mL LY900014 given SC 0-2 minutes before each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
- LY900014 Postmeal; LY900014 Postmeal-MEE: 100 U/mL LY900014 given SC 20 minutes after the start of each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Prandial insulin doses were individualized and titrated according to protocol-defined targets.
Period: Lead-in Period
Arm/Group | Insulin Lispro (Humalog) Lead-in | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog) Lead-In Maximum Extended Enrollment | Insulin Lispro (Humalog)- Maximum Extended Enrollment (MEE) | LY900014-MEE | LY900014 Postmeal-MEE
Started | 1316 | 0 | 0 | 0 | 76 | 0 | 0 | 0
Completed | 1222 | 0 | 0 | 0 | 74 | 0 | 0 | 0
Not Completed | 94 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 50 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment Interruption | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Insulin Lispro (Humalog) Lead-in | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog) Lead-In Maximum Extended Enrollment | Insulin Lispro (Humalog)- Maximum Extended Enrollment (MEE) | LY900014-MEE | LY900014 Postmeal-MEE
Started | 0 (Participants received Insulin Lispro during Lead-in Period.) | 442 (Participants were randomized to either LY900014 or Insulin lispro in Treatment Period.) | 451 (Participants were randomized to either LY900014 or Insulin lispro in Treatment Period.) | 329 (Participants were randomized to either LY900014 or Insulin lispro in Treatment Period.) | 0 (Participants received Insulin Lispro during Lead-in Period.) | 31 (Participants were randomized to either LY900014 or Insulin lispro in Treatment Period.) | 21 (Participants were randomized to either LY900014 or Insulin lispro in Treatment Period.) | 22 (Participants were randomized to either LY900014 or Insulin lispro in Treatment Period.)
Completed | 0 | 408 | 418 | 310 | 0 | 28 | 19 | 21
Not Completed | 0 | 34 | 33 | 19 | 0 | 3 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 4 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 5 | 3 | 2 | 0 | 2 | 1 | 0
Not completed — Sponsor Decision | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 20 | 23 | 14 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Insulin Lispro (Humalog)-MEE: 100 U/mL Insulin lispro given subcutaneously (SC) 0-2 minutes before each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog)-MEE | LY900014-MEE | LY900014 Postmeal-MEE | Total
Number analyzed (Participants) | 442 | 451 | 329 | 31 | 21 | 22 | 1296
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.5 (13.6) | 44.1 (13.7) | 44.5 (14.3) | 32.1 (12.3) | 32.4 (12.4) | 31.5 (12.7) | 43.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 201 | 147 | 14 | 9 | 13 | 570
  Male | 256 | 250 | 182 | 17 | 12 | 9 | 726
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 35 | 35 | 12 | 8 | 9 | 132
  Not Hispanic or Latino | 397 | 399 | 283 | 18 | 12 | 12 | 1121
  Unknown or Not Reported | 12 | 17 | 11 | 1 | 1 | 1 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 1 | 0 | 1 | 5
  Asian | 78 | 86 | 63 | 18 | 11 | 10 | 266
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 7 | 5 | 0 | 0 | 0 | 21
  White | 344 | 346 | 254 | 12 | 9 | 11 | 976
  More than one race | 11 | 10 | 5 | 0 | 1 | 0 | 27
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Argentina | 11 | 14 | 14 | 0 | 0 | 0 | 39
  Puerto Rico | 2 | 3 | 2 | 0 | 0 | 0 | 7
  Romania | 34 | 30 | 23 | 0 | 0 | 0 | 87
  United States | 129 | 134 | 98 | 0 | 0 | 0 | 361
  Japan | 59 | 62 | 46 | 0 | 0 | 0 | 167
  India | 10 | 10 | 8 | 10 | 8 | 6 | 52
  Russia | 8 | 11 | 5 | 2 | 1 | 3 | 30
  Spain | 25 | 30 | 20 | 0 | 0 | 0 | 75
  Greece | 26 | 28 | 21 | 0 | 0 | 0 | 75
  New Zealand | 10 | 11 | 3 | 0 | 0 | 0 | 24
  Austria | 9 | 6 | 7 | 0 | 0 | 0 | 22
  Sweden | 5 | 2 | 3 | 0 | 0 | 0 | 10
  Taiwan | 9 | 11 | 8 | 8 | 4 | 4 | 44
  Poland | 49 | 47 | 27 | 0 | 0 | 0 | 123
  Italy | 9 | 7 | 4 | 0 | 0 | 0 | 20
  Mexico | 6 | 4 | 8 | 11 | 8 | 9 | 46
  Slovakia | 6 | 6 | 4 | 0 | 0 | 0 | 16
  Australia | 9 | 10 | 7 | 0 | 0 | 0 | 26
  Germany | 26 | 25 | 21 | 0 | 0 | 0 | 72
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 7.33 (0.67) | 7.34 (0.65) | 7.36 (0.64) | 7.52 (0.99) | 7.28 (0.67) | 7.60 (0.62) | 7.35 (0.66)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) Efficacy Estimand at Week 26
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Least Squares (LS) mean was determined by mixed model repeated measures (MMRM) model with strata (pooled country, type of basal insulin, prandial insulin dosing plan, and HbA1c stratum) and treatment as fixed effects and baseline as a covariate. The efficacy estimand included participant data when baseline and at least one post-baseline measurement were available prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline HbA1c data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog)
Number analyzed (Participants) | 428 | 309 | 417
Percentage of HbA1c | -0.13 (0.031) | 0.08 (0.035) | -0.05 (0.031)
Statistical Analysis 1: Comparison: LY900014 vs Insulin Lispro (Humalog); Test type: Non-Inferiority — Noninferiority margin = 0.4% for HbA1c; p = 0.060, Mixed Models Analysis; LS Mean Difference = -0.08, 95% CI 2-sided [-0.16 to 0.00]
Statistical Analysis 2: Comparison: LY900014 Postmeal vs Insulin Lispro (Humalog); Test type: Non-Inferiority — Noninferiority margin = 0.4% for HbA1c; p = 0.003, Mixed Models Analysis; LS Mean Difference = 0.13, 95% CI 2-sided [0.04 to 0.22]

2. Secondary Outcome: Change From Baseline in 1-hour Postprandial Glucose (PPG) Excursion During Mixed-Meal Tolerance Test (MMTT) Efficacy Estimand at Week 26
Description: A standardized MMTT was used to characterize postprandial glucose control following administration of the study insulin. Serum glucose measured at 1-hour timepoint after the start of meal minus fasting serum glucose. 1-hour PPG excursion during MMTT uses the ANCOVA model with strata (pooled country, type of basal insulin, prandial insulin dosing plan, and HbA1c stratum) and treatment as fixed effects and baseline as a covariate. The efficacy estimand included participant data when baseline and at least one post-baseline measurement were available prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline 1-hour PPG excursion data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog)
Number analyzed (Participants) | 403 | 278 | 390
milligrams per deciliter (mg/dL) | -28.6 (3.33) | 12.5 (3.74) | -0.7 (3.34)
Statistical Analysis 1: Comparison: LY900014 vs Insulin Lispro (Humalog); Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -27.9, 95% CI 2-sided [-35.3 to -20.6]
Statistical Analysis 2: Comparison: LY900014 Postmeal vs Insulin Lispro (Humalog); Test type: Superiority; p = 0.002, ANCOVA; LS Mean Difference = 13.2, 95% CI 2-sided [5.0 to 21.4]

3. Secondary Outcome: Change From Baseline in 2-hour PPG Excursion During MMTT Efficacy Estimand at Week 26
Description: A standardized MMTT was used to characterize postprandial glucose control following administration of the study insulin. Serum glucose measured at 2-hour timepoint after the start of meal minus fasting serum glucose. 2-hour PPG excursion during MMTT uses the ANCOVA model with strata (pooled country, type of basal insulin, prandial insulin dosing plan, and HbA1c stratum) and treatment as fixed effects and baseline as a covariate. The efficacy estimand included participant data when baseline and at least one post-baseline measurement were available prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline 2-hour PPG excursion data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog)
Number analyzed (Participants) | 401 | 278 | 391
mg/dL | -34.7 (4.50) | -10.2 (5.04) | -3.5 (4.51)
Statistical Analysis 1: Comparison: LY900014 vs Insulin Lispro (Humalog); Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -31.2, 95% CI 2-sided [-41.1 to -21.2]
Statistical Analysis 2: Comparison: LY900014 Postmeal vs Insulin Lispro (Humalog); Test type: Superiority; p = 0.235, ANCOVA; LS Mean Difference = -6.7, 95% CI 2-sided [-17.6 to 4.3]

4. Secondary Outcome: Rate of Severe Hypoglycemia at Week 26
Description: Severe hypoglycemia is defined as an event requiring assistance of another person to administer carbohydrate, glucagon, or other resuscitative actions. During these episodes, the participant has an altered mental status and cannot assist in his or her own care, or may be semiconscious or unconscious, or experience coma with or without seizures, and may require parenteral therapy. Rate of severe hypoglycemia events per 100 years during a defined period was calculated by total number of severe hypoglycemia episodes within the period divided by the cumulative days on treatment from all participants within a treatment group *36525.
Time Frame: Baseline through Week 26
Population: All randomized participants with evaluable hypoglycemic data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: Events per 100 participant years
Arm/Group | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog)
Number analyzed (Participants) | 451 | 329 | 442
Events per 100 participant years | 16.50 | 13.70 | 18.34

5. Secondary Outcome: Rate of Documented Symptomatic Hypoglycemia at Week 26
Description: Documented symptomatic hypoglycemia is an event during which typical symptoms of hypoglycemia are accompanied by blood glucose (BG) of <54 mg/dL [3.0 millimole per liter (mmol/L)]. The rate of documented symptomatic hypoglycemia was estimated by negative binomial model: number of episodes = treatment with log (treatment exposure in days/365.25) as an offset variable.
Time Frame: Baseline through Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Events per participant per year
Arm/Group | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog)
Number analyzed (Participants) | 451 | 329 | 442
Events per participant per year | 6.71 (0.479) | 7.75 (0.582) | 7.35 (0.697)

6. Secondary Outcome: Change From Baseline in 1,5-Anhydroglucitol (1,5-AG) at Week 26
Description: 1,5-anhydroglucitol (1,5-AG) is a marker of short-term glycemic control especially postprandial hyperglycemia. 1,5-AG accurately predicts rapid changes in glycemia and is tightly associated with glucose fluctuations and postprandial glucose. LS Mean was calculated using mixed model repeated measures (MMRM) including fixed class effects of treatment, strata (pooled country, type of basal insulin, HbA1c stratum and number of prandial doses at study entry), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline value. The analysis included data collected prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline 1,5-AG data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: milligram per liter (mg/L)
Arm/Group | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog)
Number analyzed (Participants) | 430 | 307 | 417
milligram per liter (mg/L) | 0.19 (0.108) | -0.38 (0.124) | -0.22 (0.109)

7. Secondary Outcome: Change From Baseline in 10-Point Self-Monitoring Blood Glucose (SMBG) Values at Week 26
Description: SMBG 10-point profiles were measured at fasting, 1-hour post morning meal, 2-hours post morning meal, pre midday meal, 1-hour post midday meal, 2-hours post midday meal, pre evening meal, 1-hour post evening meal, 2-hours post evening meal, and bedtime. LS Mean was analyzed using mixed model repeated measures (MMRM) including fixed class effects of treatment, strata (pooled country, type of basal insulin, HbA1c stratum and number of prandial doses at study entry), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline value. The efficacy estimand included participant data when baseline and at least one post-baseline measurement prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline SMBG data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog)
Number analyzed (Participants) | 314 | 230 | 300
mg/dL
  Morning Premeal: number analyzed (Participants) | 310 | 230 | 300
  Morning Premeal | -1.1 (2.82) | 2.9 (3.19) | -3.3 (2.84)
  Morning 1-hour Postmeal: number analyzed (Participants) | 294 | 218 | 282
  Morning 1-hour Postmeal | -14.8 (3.30) | 5.4 (3.71) | -1.0 (3.31)
  Morning 2-hour Postmeal: number analyzed (Participants) | 300 | 221 | 292
  Morning 2-hour Postmeal | -10.1 (3.21) | -0.2 (3.63) | 1.4 (3.22)
  Midday Premeal: number analyzed (Participants) | 314 | 230 | 298
  Midday Premeal | 6.6 (2.80) | 4.0 (3.17) | 1.9 (2.83)
  Midday 1-hour Postmeal: number analyzed (Participants) | 295 | 216 | 280
  Midday 1-hour Postmeal | -2.2 (3.36) | 11.4 (3.81) | 1.4 (3.40)
  Midday 2-hour Postmeal: number analyzed (Participants) | 300 | 221 | 288
  Midday 2-hour Postmeal | -5.2 (3.24) | 0.0 (3.67) | -2.7 (3.28)
  Evening Premeal: number analyzed (Participants) | 313 | 228 | 298
  Evening Premeal | 5.2 (3.21) | 0.4 (3.64) | -1.4 (3.24)
  Evening 1-hour Postmeal: number analyzed (Participants) | 290 | 218 | 278
  Evening 1-hour Postmeal | -7.0 (3.53) | 15.3 (3.95) | -0.9 (3.57)
  Evening 2-hour Postmeal: number analyzed (Participants) | 292 | 217 | 278
  Evening 2-hour Postmeal | -8.2 (3.43) | -1.6 (3.83) | -0.6 (3.45)
  Bedtime: number analyzed (Participants) | 276 | 196 | 272
  Bedtime | -6.8 (3.58) | -11.0 (4.08) | -2.9 (3.56)

8. Secondary Outcome: Change From Baseline in Insulin Dose at Week 26
Description: LS Mean was analyzed using mixed model repeated measures (MMRM) including fixed class effects of treatment, strata (pooled country, type of basal insulin, HbA1c stratum and number of prandial doses at study entry), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline value. The analysis included data prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline basal insulin dose data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: Units (U)/day
Arm/Group | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog)
Number analyzed (Participants) | 400 | 285 | 379
Units (U)/day
  Total Daily Insulin Dose: number analyzed (Participants) | 388 | 278 | 367
  Total Daily Insulin Dose | 2.9 (0.72) | 2.2 (0.83) | 2.0 (0.73)
  Daily Basal Insulin Dose: number analyzed (Participants) | 390 | 283 | 371
  Daily Basal Insulin Dose | 1.0 (0.28) | 1.2 (0.33) | 0.9 (0.29)
  Daily Prandial Insulin Dose | 1.5 (0.59) | 1.0 (0.68) | 0.9 (0.60)

9. Secondary Outcome: Change From Baseline in Insulin Treatment Satisfaction Questionnaire (ITSQ) Regimen Inconvenience Domain Score at Week 26
Description: ITSQ is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. The questionnaire measures satisfaction from the following 5 domains: Inconvenience of Regimen, Lifestyle Flexibility, Glycemic Control, Hypoglycemic Control, and Insulin Delivery Device. Data presented are the transformed overall score on a scale of 0-100, where higher scores indicate better treatment satisfaction. LS Mean was calculated using the ANCOVA model with strata (pooled country, type of basal insulin, number of prandial doses at study entry, and HbA1c stratum), and treatment as fixed effects and baseline as covariate. The analysis included data prior to permanent discontinuation of study drug. The analysis included data prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and post-baseline data. Missing endpoints were imputed by applying the Last Observation Carried Forward (LOCF) method to post-baseline data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog)
Number analyzed (Participants) | 432 | 314 | 423
Units on a scale | 1.4 (0.92) | 1.5 (1.01) | 0.7 (0.91)

10. Secondary Outcome: Change From Baseline in ITSQ Lifestyle Flexibility Domain Score at Week 26
Description: ITSQ is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. The questionnaire measures satisfaction from the following 5 domains: Inconvenience of Regimen, Lifestyle Flexibility, Glycemic Control, Hypoglycemic Control, and Insulin Delivery Device. Data presented are the transformed overall score on a scale of 0-100, where higher scores indicate better treatment satisfaction. LS Mean was calculated using the analysis of covariance (ANCOVA) with strata (pooled country, type of basal insulin, number of prandial doses at study entry, and HbA1c stratum), and treatment as fixed effects and baseline as covariate. The analysis included data prior to permanent discontinuation of study drug. The analysis included data prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and post-baseline data. Missing endpoints were imputed by applying the LOCF method to the post-baseline data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog)
Number analyzed (Participants) | 432 | 314 | 423
Units on a scale | 2.1 (1.09) | 3.7 (1.19) | 1.3 (1.07)

11. Secondary Outcome: Percentage of Participants With HbA1c <7%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 26
Population: All randomized participants with baseline and at least one post-baseline HbA1c <7% data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: Percentage of participants
Arm/Group | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog)
Number analyzed (Participants) | 450 | 322 | 442
Percentage of participants | 36.00 | 24.84 | 33.94

12. Secondary Outcome: Change From Baseline in HbA1c at Week 52
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Least Squares (LS) mean was determined by MMRM model with variables of baseline, pooled country, type of basal insulin during lead-in, prandial Insulin Dosing Plan, treatment (Type III sum of squares) as fixed factors. The analysis included data prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 52
Population: All randomized participants with baseline and at least one postbaseline observation for HbA1c. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups. Only double blind arms analysed for this outcome because open label group ended at week 26.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | LY900014 | Insulin Lispro (Humalog)
Number analyzed (Participants) | 410 | 400
Percentage of HbA1c | 0.13 (0.036) | 0.20 (0.037)
Statistical Analysis 1: Comparison: LY900014 vs Insulin Lispro (Humalog); Test type: Superiority; p = 0.184, Mixed Models Analysis; LS Mean Difference = -0.06, 95% CI 2-sided [-0.16 to 0.03]

ADVERSE EVENTS:
Time Frame: Up to 56 Weeks
Description: All randomized participants. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Groups:
- Insulin Lispro (Humalog) Lead-in; Insulin Lispro (Humalog); Insulin Lispro (Humalog) Lead-in-MEE; Insulin Lispro (Humalog)-MEE: 100 U/mL Insulin lispro given subcutaneously (SC) 0-2 minutes before each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
Arm/Group | Insulin Lispro (Humalog) Lead-in | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal | Insulin Lispro (Humalog) Lead-in-MEE | Insulin Lispro (Humalog)-MEE | LY900014-MEE | LY900014 Postmeal-MEE
All-Cause Mortality (participants affected / at risk) | 0/1316 | 1/442 | 1/451 | 1/329 | 0/76 | 0/31 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 48/1316 | 67/442 | 54/451 | 30/329 | 0/76 | 9/31 | 3/21 | 2/22
Other Adverse Events (participants affected / at risk) | 131/1316 | 147/442 | 163/451 | 104/329 | 5/76 | 13/31 | 3/21 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Lispro (Humalog) Lead-in (N=1316) | Insulin Lispro (Humalog) (N=442) | LY900014 (N=451) | LY900014 Postmeal (N=329) | Insulin Lispro (Humalog) Lead-in-MEE (N=76) | Insulin Lispro (Humalog)-MEE (N=31) | LY900014-MEE (N=21) | LY900014 Postmeal-MEE (N=22)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0/743 (0) | 1/256 (1) | 0/250 (0) | 0/182 (0) | 0/40 (0) | 0/17 (0) | 0/12 (0) | 0/9 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urogenital infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pericarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brachial plexus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 33 (38) | 39 (69) | 33 (52) | 16 (23) | 0 (0) | 3 (5) | 3 (6) | 2 (3)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dural arteriovenous fistula (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0/573 (0) | 0/186 (0) | 0/201 (0) | 1/147 (1) | 0/36 (0) | 0/14 (0) | 0/9 (0) | 0/13 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/573 (0) | 0/186 (0) | 1/201 (1) | 1/147 (1) | 0/36 (0) | 0/14 (0) | 0/9 (0) | 0/13 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/573 (0) | 0/186 (0) | 1/201 (1) | 0/147 (0) | 0/36 (0) | 0/14 (0) | 0/9 (0) | 0/13 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0/573 (0) | 1/186 (1) | 0/201 (0) | 0/147 (0) | 0/36 (0) | 0/14 (0) | 0/9 (0) | 0/13 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0/573 (0) | 1/186 (1) | 0/201 (0) | 0/147 (0) | 0/36 (0) | 0/14 (0) | 0/9 (0) | 0/13 (0)
Uterine polyp (Reproductive system and breast disorders) | 0/573 (0) | 0/186 (0) | 1/201 (1) | 0/147 (0) | 0/36 (0) | 0/14 (0) | 0/9 (0) | 0/13 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Lispro (Humalog) Lead-in (N=1316) | Insulin Lispro (Humalog) (N=442) | LY900014 (N=451) | LY900014 Postmeal (N=329) | Insulin Lispro (Humalog) Lead-in-MEE (N=76) | Insulin Lispro (Humalog)-MEE (N=31) | LY900014-MEE (N=21) | LY900014 Postmeal-MEE (N=22)
Pyrexia (General disorders) | 4 (4) | 2 (2) | 6 (7) | 8 (8) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 24 (24) | 24 (25) | 15 (16) | 1 (1) | 3 (4) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 85 (87) | 88 (123) | 106 (161) | 66 (85) | 1 (1) | 5 (7) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 3 (3) | 4 (5) | 6 (6) | 4 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 25 (25) | 33 (43) | 28 (34) | 19 (22) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 2/573 (2) | 3/186 (3) | 2/201 (2) | 2/147 (2) | 0/36 (0) | 1/14 (1) | 0/9 (0) | 0/13 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 4 (5) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0/573 (0) | 0/186 (0) | 0/201 (0) | 0/147 (0) | 0/36 (0) | 1/14 (1) | 0/9 (0) | 0/13 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0/573 (0) | 0/186 (0) | 0/201 (0) | 0/147 (0) | 0/36 (0) | 1/14 (1) | 0/9 (0) | 0/13 (0)
Retroplacental haematoma (Pregnancy, puerperium and perinatal conditions) | 0/573 (0) | 0/186 (0) | 0/201 (0) | 0/147 (0) | 0/36 (0) | 1/14 (1) | 0/9 (0) | 0/13 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/573 (1) | 0/186 (0) | 1/201 (1) | 0/147 (0) | 0/36 (0) | 1/14 (1) | 0/9 (0) | 0/13 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (5) | 7 (7) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vasectomy (Surgical and medical procedures) | 0/743 (0) | 0/256 (0) | 0/250 (0) | 0/182 (0) | 0/40 (0) | 1/17 (1) | 0/12 (0) | 0/9 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT03214367/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT03214367/SAP_001.pdf